CLINICAL TRIAL: NCT05656443
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase Ⅱ/Ⅲ Clinical Study to Evaluate the Efficacy and Safety of GST-HG171/Ritonavir in Patients With Mild to Moderate COVID-19
Brief Title: Study of GST-HG171/Ritonavir Compared With Placebo in Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GST-HG171-II/III-01
Record Dates: First submitted 2022-12-16; First posted 2022-12-19 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GST-HG171/Ritonavir (Experimental)
  Interventions: Drug: GST-HG171/Ritonavir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GST-HG171/Ritonavir — dose of 150 mg GST-HG171 with 100 mg ritonavir
  Arms: GST-HG171/Ritonavir
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled clinical trial to assess the efficacy and safety of GST-HG171/Ritonavir in the treatment of mild to moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years when signing the informed consent form (ICF);
2. Subjects with reverse transcription-polymerase chain reaction (RT-PCR) test positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in specimens such as nasopharyngeal swabs/oropharyngeal swabs for the first time within 4 days prior to randomization who meet the diagnostic and treatment criteria for mild and moderate cases in the Diagnosis and Treatment Protocol for COVID-19 (Trial Version 9) issued by the National Health Commission of the Peoples Republic of China ;
3. RT-PCR result of N gene or ORF gene of SARS-CoV-2 within 48 hours before randomization shows a Ct value < 35; at least 2 COVID-19 target symptoms appeared for the first time within 72 hours before randomization (COVID-19 target symptoms include fever, cough, stuffy or runny nose, sore throat or dry throat, shortness of breath or difficulty breathing, headache, muscle or body aches, diarrhoea, chills, nausea, and vomit), including at least one designated symptom: fever, cough, stuffy or runny nose, sore throat or dry throat, shortness of breath or difficulty breathing;
4. Women of childbearing potential must have a negative serum pregnancy test during the screening period. Subjects should take effective contraceptive measures throughout the study period since signing the informed consent form and for 28 days after the end of the study;
5. Subjects who are able to understand the study procedures and methods, and voluntarily participate in the study and sign the ICF after being fully informed.

Exclusion Criteria:

1. Subjects who are known to have hypersensitivity to any component of the investigational drug;
2. Subjects who meet diagnostic and treatment criteria for severe and critical cases in the Diagnosis and Treatment Protocol for COVID-19 (Trial Version 10) issued by National Health Commission of the People's Republic of China;
3. Abnormal hepatic function at screening: total bilirubin ≥ 1.5 × upper limit of normal (ULN); ALT or AST ≥ 3 × ULN;
4. Human immunodeficiency virus (HIV) antibody positive, treponema pallidum-specific antibody (TP-PA) positive or rapid plasma reagin (RPR) positive for syphilis at screening;
5. Abnormal renal function at screening: serum creatinine ≥ 1.5 × ULN;
6. Subjects with impaired immune system (including those treated with corticosteroids* or other immunosuppressants*, or those with progression or recurrence of cancer) at screening; Note: *Patients using skin preparations are allowed to be enrolled, but the skin preparations cannot be used in the eyes, nose or ears or by inhalation.
7. Acute onset of chronic respiratory diseases, including bronchial asthma and chronic obstructive pulmonary disease at screening;
8. There are suspected or confirmed acute systemic infections except for COVID-19 at the time of screening (for example, the pathogen detection indicates that it is complicated with influenza; there is a high possibility of bacterial infection as indicated by symptoms, signs, laboratory tests or imaging), which may interfere with the assessment of response to study intervention;
9. Any comorbidity requiring surgery within 14 days prior to randomization or during the study, or any life-threatening comorbidity within 30 days prior to randomization as determined by the investigator;
10. Subjects who are receiving HIV antiviral treatment at screening;
11. Treatment with SARS-CoV-2 antiviral drugs within 14 days prior to randomization;
12. Subjects who have received (within 30 days prior to randomization or within 5 drug half-lives, whichever is longer) or are expected to receive COVID-19 monoclonal antibody, intravenous injection of COVID-19 human immunoglobulin, or COVID-19 convalescent plasma therapy;
13. Subjects who have received any COVID-19 vaccine within 28 days prior to randomization or planned to receive any COVID-19 vaccine during the study;
14. Any drug prohibited by the package insert of Paxlovid that is currently used or expected to be used during treatment and within 4 days after the last dose of study drug, or any other drug or substance that is highly dependent on cytochrome P450 (CYP) 3A4, CYP2B6, CYP1A2, multidrug resistance gene 1 (MDR1) or organic anion transporting polypeptide (OATP) 1B3 for clearance; any potent CYP3A4 or MDR1 inducers used within 28 days prior to randomization or expected to be used during treatment and within 4 days after the last dose of study drug ;
15. Pregnant or lactating women;
16. Subjects who have participated in other clinical trials within 3 months prior to administration or are receiving other investigational drugs;
17. Subjects with other conditions that, in the judgment of the investigator, make them unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Time to sustained clinical recovery of 11 COVID-19 symptoms | Day 1 through Day 28
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 for two consecutive days

SECONDARY OUTCOMES:
Viral load | Baseline through Day 5
  Change of viral load compared to the baseline
Time to sustained clinical recovery of 5 COVID-19 symptoms | Day 1 through Day 28
  The time from the start of treatment to the time when respiratory and feverish symptoms get scores of 0 for two consecutive days
Time to sustained alleviation of 11 COVID-19 symptoms | Baseline through Day 28
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 or 1 for two consecutive days
Proportion of participants in clinical recovery | Day 1 through Day 28
  Proportion of participants in clinical recovery
AE | Day 1 through Day 28
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lu H, Zhang G, Mao J, Chen X, Zhan Y, Lin L, Zhang T, Tang Y, Lin F, Zhu F, Lin Y, Zeng Y, Zhang K, Yuan W, Liang Z, Sun R, Huo L, Hu P, Lin Y, Zhuang X, Wei Z, Chen X, Yan W, Yan X, Mu L, Lin Z, Tu X, Tan H, Huang F, Hu Z, Li H, Li G, Fu H, Yang Z, Chen X, Wang FS, Zhong N. Efficacy and safety of GST-HG171 in adult patients with mild to moderate COVID-19: a randomised, double-blind, placebo-controlled phase 2/3 trial. EClinicalMedicine. 2024 Apr 10;71:102582. doi: 10.1016/j.eclinm.2024.102582. eCollection 2024 May. PMID 38618202